CLINICAL TRIAL: NCT00886639
Title: Effect Of Oxygen-Supply On The 6-Minute-Walking-Distance in Patients With Chronic Obstructive Pulmonary Disease (COPD) GOLD Stage III/IV Before And After A Multimodal Rehabilitation
Brief Title: Effect of Oxygen-supply on 6-Minute-Walking-Distance of COPD III/IV-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: ROX Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: BGL O2
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD III/IV; Oxygen Supply; Six-Minute-Walking-Test; Oxygen Responder
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- First of 2 6-minute-walking test with oxygen (Other): Continuous flow of 2 liters per minute First with oxygen, second with medical air
  Interventions: Other: 6MWT with oxygen; Other: 6MWT with medical air
- First of 2 6-minute-walking tests with medical air (Other): Medical air is compressed room air. First test with medical air, second with oxygen
  Interventions: Other: 6MWT with oxygen; Other: 6MWT with medical air

INTERVENTIONS:
Other: 6MWT with oxygen — 2 liter per minute as continuous-flow
Other: 6MWT with medical air — 2 liters as continuous-flow

SUMMARY:
The aim of this study is to investigate the six-minute-walking-distance of COPD-patients with breathing oxygen in comparison to breathing normal air. Patients, who increase their walking-distance about more than 15% or 35m only because of breathing oxygen, are so-called "Oxygen Responders." The study is aimed to find attributes of Oxygen Responder and to investigate, if a patient can change the "respond" with higher performance and endurance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease III/IV

Exclusion Criteria:

* Severe exacerbations in the last 4 weeks prior to begin of study (definition of exacerbation: symptoms on more than 3 days with a relevant change in drug therapy (cortisone, antibiotics))
* Severe exacerbation during rehabilitation
* Cardiac insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Dr.med., Study Director — Klinikum Berchtesgadener Land, Schön Kliniken; Inga Heinzelmann, Dipl. Sportw, Principal Investigator — Klinikum Berchtesgadener Land, Schön Kliniken
Locations (1):
- Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee, Germany

REFERENCES:
- [Derived] Jarosch I, Gloeckl R, Damm E, Schwedhelm AL, Buhrow D, Jerrentrup A, Spruit MA, Kenn K. Short-term Effects of Supplemental Oxygen on 6-Min Walk Test Outcomes in Patients With COPD: A Randomized, Placebo-Controlled, Single-blind, Crossover Trial. Chest. 2017 Apr;151(4):795-803. doi: 10.1016/j.chest.2016.11.044. Epub 2016 Dec 8. PMID 27940278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: inpatient rehabilitation programme, recruitment directly after admission.
Period: Overall Study
Arm/Group | 6MWT With Different Gas Mixtures
Started | 127
Completed | 111
Not Completed | 16
Not completed — acute exacerbation | 14
Not completed — non-compliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | 6MWT With Different Gas Mixtures
Number analyzed (Participants) | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 67
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 73
Region of Enrollment [Number; unit: participants]
  Germany | 127
Forced expiratory volume in 1 second (FEV1%pred.) [Mean (Standard Deviation); unit: percentage of predicted value] — in percentage of predicted value
  percentage of predicted value | 35.5 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Response
Description: Change in oxygen response (6-minute-walking distance on oxygen minus 6-minute-walking distance on medical air) from baseline to 3 weeks
Time Frame: day 1 and day 2; day 21 and day 22
Population: per protocol
Measure: Mean (Standard Deviation); unit: Meter
Groups:
- Oxygen Response: difference between 6-minute-walking test on oxygen and on medical air
Arm/Group | Oxygen Response
Number analyzed (Participants) | 111
Meter | 26.9 (41.9)

2. Secondary Outcome: Oxygen Partial Pressure (paO2)
Description: change in paO2 from minute 0 to minute 6 in 6-minute-walking test on oxygen/ medical air
Time Frame: day 1: minute "0" and "6"
Reporting Status: Not Posted

3. Secondary Outcome: Diffusion Capacity
Description: change in diffusion capacity from baseline to 3 weeks
Time Frame: day 1 and 21
Reporting Status: Not Posted

4. Secondary Outcome: Lung Function
Description: change in lung function from baseline to 3 weeks
Time Frame: day 1 and 21
Reporting Status: Not Posted

5. Secondary Outcome: BORG-Score
Description: change of BORG-Score from pre to post 6 minute-walking test (minute 0 and 6)on oxygen/ medical air
Time Frame: day 1: minute 0 and minute 6
Reporting Status: Not Posted

6. Secondary Outcome: Oxygen Saturation
Description: Change of oxygen saturation from minute 0 to 6 in 6Minute-walking test on oxygen/ medical air
Time Frame: day 1: minute 0 and 6
Reporting Status: Not Posted

7. Secondary Outcome: Oxygen Partial Pressure (paO2)
Description: change in paO2 from minute 0 to minute 6 in 6-minute-walking test on oxygen/ medical air
Time Frame: day 21: minute 0 and minute 6
Reporting Status: Not Posted

8. Secondary Outcome: BORG-Score
Description: change of BORG-Score from pre to post 6 minute-walking test (minute 0 and 6)on oxygen/ medical air
Time Frame: day 2: minute 0 and minute 6
Reporting Status: Not Posted

9. Secondary Outcome: BORG-Score
Description: change of BORG-Score from pre to post 6 minute-walking test (minute 0 and 6)on oxygen/ medical air
Time Frame: day 22: minute 0 and minute 6
Reporting Status: Not Posted

10. Secondary Outcome: BORG-Score
Description: change of BORG-Score from pre to post 6 minute-walking test (minute 0 and 6)on oxygen/ medical air
Time Frame: day 21: minute 0 and minute 6
Reporting Status: Not Posted

11. Secondary Outcome: Oxygen Partial Pressure (paO2)
Description: change in paO2 from minute 0 to minute 6 in 6-minute-walking test on oxygen/ medical air
Time Frame: day 20: minute 0 and minute 6
Reporting Status: Not Posted

12. Secondary Outcome: Oxygen Partial Pressure (paO2)
Description: change in paO2 from minute 0 to minute 6 in 6-minute-walking test on oxygen/ medical air
Time Frame: day 2: minute "0" and "6"
Reporting Status: Not Posted

13. Secondary Outcome: Oxygen Saturation
Description: Change of oxygen saturation from minute 0 to 6 in 6Minute-walking test on oxygen/ medical air
Time Frame: day 2: minute 0 and 6
Reporting Status: Not Posted

14. Secondary Outcome: Oxygen Saturation
Description: Change of oxygen saturation from minute 0 to 6 in 6Minute-walking test on oxygen/ medical air
Time Frame: day 21: minute 0 and 6
Reporting Status: Not Posted

15. Secondary Outcome: Oxygen Saturation
Description: Change of oxygen saturation from minute 0 to 6 in 6Minute-walking test on oxygen/ medical air
Time Frame: day 22: minute 0 and 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 6MWT With Different Gas Mixtures
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes